CLINICAL TRIAL: NCT01358045
Title: Topical Vitamin D3, Diclofenac or a Combination of Both to Treat Basal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEC 10-2-088
Record Dates: First submitted 2011-05-17; First posted 2011-05-23 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Basal Cell Carcinoma
Keywords: Topical; Diclofenac; Vitamin D3
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Diclofenac; Calcitriol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Solaraze (Active Comparator)
  Interventions: Drug: Diclofenac
- Solaraze + Silkis (Active Comparator)
  Interventions: Drug: Diclofenac + Calcitriol
- Silkis (Active Comparator)
  Interventions: Drug: Calcitriol
- No treatment (No Intervention)

INTERVENTIONS:
Drug: Diclofenac — Application on the lesion 2 times a day 8 weeks.
  Other Names: Solaraze
  Arms: Solaraze
Drug: Diclofenac + Calcitriol — Application on the lesion 2 times a day, both ointments, 8 weeks.
  Other Names: Solaraze + Silkis
  Arms: Solaraze + Silkis
Drug: Calcitriol — Application on the lesion, 2 times a day, 8 weeks.
  Other Names: Silkis
  Arms: Silkis

SUMMARY:
Basal cell carcinoma (BCC) is the most frequent malignant tumor in Caucasians and the incidence is still increasing with 3-8% each year. Since BCCs generally occur on sun-exposed areas of the skin, the rice in incidence is mainly explained by the increasing exposure to (intermittent) ultraviolet radiation. Surgical excision is still the standard treatment for (micro)nodular BCCs. The costs as well as the increased workload are stressing the health care system even further and posing BCC an important health care problem. Since half of the BCCs arise primarily on the face & (bald) head and treatment by surgical excision may result in disfiguring scars, patients often experience a dramatic decrease of their quality of life. Hence, there is an urgent medical and societal need for a simple and cheap (targeted) treatment, preferably to be performed by the patients themselves. This treatment must be safe and effective. Such treatment is not available yet. BCC tumorigenesis is complex and must be multifactorial. Genetic alterations of multiple components of the Sonic Hedgehog (SHH) pathway are involved in sporadic BCC pathogenesis; inactivating mutations in Patched-1 (PTCH1) and activating mutations of Smoothened (SMO) and Suppressor of Fused (SU(FU)). With this knowledge, inhibition of the SHH pathway by SMO antagonists was successfully administered, however treatment resulted only in partial clinical response ofBCC. Recently, involvement of the Wingless (Wnt) pathway has been proven to be essential in BCC tumorigenic response. Moreover, a recent study of our own department provides the first evidence that epigenetic alterations, particularly promoter hypermethylation, influence both the SHH and Wnt pathway (own data, not published), which can serve as therapeutic targets. Both non-steroidal anti-inflammatory drugs (NSAlDS) and vitamin D derivatives are able to directly or indirectly target the Wnt pathway. Furthermore, vitamin D3 is able to inhibit Smoothened (SMO) in vitro, resulting in inhibition of the SHH pathway. Although in vivo studies are lacking, the investigators assume that topical application of these drugs may inhibit BCC growth and/or may cure BCC and thus might provide very promising future perspectives. Calcitriol and NSAlDs ointments are both already available for other indications and save in use. Eventually, our approach may result in a systematic approach to BCC, targeting (epi)genetic changes to treat and/or prevent further tumour growth.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 18 years
* Primary basal cell carcinoma, histologically confirmed
* (Micro) Nodular or superficial histological subtype
* Comorbidities may not interfere with study treatment
* Capable to understand instructions

Exclusion Criteria:

* Age under 18 years
* Tumors located at the H-zone of the face
* Deficient histological conformation
* Proven or suspected malignancy of other organs
* Not capable of comprehending instructions
* Incompetent
* Use of oral NSAlDs during the trial period or within 30 days before starting therapy
* Use of oral vitamin D (containing) supplements during the trial period or within 30 days before starting therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-11; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Histological changes in different proliferation and apoptosis markers. | At baseline and after 8 weeks.
  To determine the change in mean percentage of cells expressing Ki67 and BCL2 after topical application of Calcitriol (Silkis) 3 μg/g, Diclofenac 3% or a combination of both.

SECONDARY OUTCOMES:
Macroscopic tumour changes | Baseline and after 8 weeks.
  We want the observe if the tumour will also macroscopically change within 8 weeks of treatment. Things were we will focus on will be size and colour.
Toleration | 8 weeks
  We want to evaluate if the patients will tolerate the therapy. Main points in here will be irritation of the skin and the amount of time this therapy costs the patients.
Compliance | 8 weeks
  Data for compliance with the prescribed regimens of either diclofenac sodium-3% gel, calcitriol 3µg/g ointment or a combination of both will be obtained from a personal diary kept by patients and completed once a week during treatment. Compliance was calculated as the number of applications done by the patient divided by the total prescribed number of applications.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands